CLINICAL TRIAL: NCT00680017
Title: A 30-Week, Multicenter, Randomized, Double-Blind, Parallel-Group Study of the Combination of ABT-335 and Rosuvastatin Compared to Rosuvastatin Monotherapy in Dyslipidemic Subjects With Stage 3 Chronic Kidney Disease
Brief Title: 30 Week Study of the Combination of ABT-335 and Rosuvastatin Compared to Rosuvastatin Monotherapy for Subjects With Dyslipidemia and Stage 3 Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-313
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Dyslipidemia; Kidney Disease
Keywords: Dyslipidemia; Kidney Disease
MeSH Terms: conditions — Dyslipidemias; Kidney Diseases | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium; fenofibric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ABT-335 plus rosuvastatin (Experimental): ABT-335 45 mg plus rosuvastatin 5 mg for 8 weeks, then ABT-335 45 mg plus rosuvastatin 10 mg for 8 weeks
  Interventions: Drug: ABT-335 plus rosuvastatin
- Rosuvastatin (Active Comparator): Rosuvastatin 5 mg for 8 weeks then rosuvastatin 10 mg for 8 weeks
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: ABT-335 plus rosuvastatin — ABT-335 45 mg plus rosuvastatin 5 mg for 8 weeks, then ABT-335 45 mg plus rosuvastatin 10 mg for 8 weeks
  Other Names: fenofibric acid and rosuvastatin
  Arms: ABT-335 plus rosuvastatin
Drug: Rosuvastatin — Rosuvastatin 5 mg for 8 weeks then rosuvastatin 10 mg for 8 weeks
  Other Names: rosuvastatin, Crestor
  Arms: Rosuvastatin

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the combination of ABT-335 plus rosuvastatin in dyslipidemic subjects with Chronic Kidney Disease (CKD) Stage 3.

ELIGIBILITY:
Inclusion Criteria

* Dyslipidemic participants with Chronic Kidney Disease Stage 3
* For entry into the Treatment Phase (Visit 3), the participant satisfied the following laboratory criteria (measured at the Screening Visit[s]):

  * Estimated glomerular filtration rate between 30 and 59 mL/min/1.73 m2 (Chronic Kidney Disease Stage 3) by simplified 4 variable Modification of Diet in Renal Disease formula (this includes a 10 percent variation in the upper limit of estimated glomerular filtration rate that was allowed for the enrollment of participants to account for variability in the creatinine assay).
  * Fasting lipid results following greater than or equal to 12-hour fasting period:
* Triglycerides level greater than or equal to 150 mg/dL,
* High-density lipoprotein cholesterol less than 40 mg/dL for males and less than 50 mg/dL for females, and
* Low-density lipoprotein cholesterol greater than or equal to 130 mg/dL Exclusion Criteria
* Participants with certain chronic or unstable medical conditions.
* Participants with unstable dose of medications or receiving coumarin anticoagulants, systemic cyclosporine, or certain other medications.
* Pregnant or lactating women, or women intending to become pregnant.
* Participants with diabetes mellitus that is poorly controlled.
* Participants of Asian ancestry (having Filipino, Chinese, Japanese, Korean, Vietnamese, or Asian-Indian origin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (114):
- United States (102):
  - Site Reference ID/Investigator# 22521, Birmingham, Alabama
  - Site Reference ID/Investigator# 22478, Huntsville, Alabama
  - Site Reference ID/Investigator# 8365, Madison, Alabama
  - Site Reference ID/Investigator# 8416, Montgomery, Alabama
  - Site Reference ID/Investigator# 7869, Chula Vista, California
  - Site Reference ID/Investigator# 8435, Fountain Valley, California
  - Site Reference ID/Investigator# 22487, Lincoln, California
  - Site Reference ID/Investigator# 22426, Long Beach, California
  - Site Reference ID/Investigator# 8096, Los Angeles, California
  - Site Reference ID/Investigator# 22962, Norwalk, California
  - Site Reference ID/Investigator# 8311, Riverside, California
  - Site Reference ID/Investigator# 22816, Sacramento, California
  - Site Reference ID/Investigator# 8510, Simi Valley, California
  - Site Reference ID/Investigator# 22821, West Hills, California
  - Site Reference ID/Investigator# 7958, Arvada, Colorado
  - Site Reference ID/Investigator# 15881, Denver, Colorado
  - Site Reference ID/Investigator# 8399, Westminster, Colorado
  - Site Reference ID/Investigator# 23224, Boynton Beach, Florida
  - Site Reference ID/Investigator# 22474, Clearwater, Florida
  - Site Reference ID/Investigator# 21803, Coral Springs, Florida
  - Site Reference ID/Investigator# 22811, Daytona Beach, Florida
  - Site Reference ID/Investigator# 27103, Hollywood, Florida
  - Site Reference ID/Investigator# 8398, Hudson, Florida
  - Site Reference ID/Investigator# 26723, Kissimmee, Florida
  - Site Reference ID/Investigator# 37676, Kissimmee, Florida
  - Site Reference ID/Investigator# 8231, Lauderdale Lakes, Florida
  - Site Reference ID/Investigator# 22486, Longwood, Florida
  - Site Reference ID/Investigator# 22520, New Port Richey, Florida
  - Site Reference ID/Investigator# 8226, Orlando, Florida
  - Site Reference ID/Investigator# 22477, Ormond Beach, Florida
  - Site Reference ID/Investigator# 8386, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 22518, Plant City, Florida
  - Site Reference ID/Investigator# 12882, Port Charlotte, Florida
  - Site Reference ID/Investigator# 37675, Saint Cloud, Florida
  - Site Reference ID/Investigator# 8410, West Palm Beach, Florida
  - Site Reference ID/Investigator# 21802, Winter Haven, Florida
  - Site Reference ID/Investigator# 8136, Atlanta, Georgia
  - Site Reference ID/Investigator# 23503, Dunwoody, Georgia
  - Site Reference ID/Investigator# 7948, Macon, Georgia
  - Site Reference ID/Investigator# 22819, Roswell, Georgia
  - Site Reference ID/Investigator# 22813, Suwanee, Georgia
  - Site Reference ID/Investigator# 27682, Chicago, Illinois
  - Site Reference ID/Investigator# 8227, Peoria, Illinois
  - Site Reference ID/Investigator# 13922, Mishawaka, Indiana
  - Site Reference ID/Investigator# 8094, Council Bluffs, Iowa
  - Site Reference ID/Investigator# 22430, Iowa City, Iowa
  - Site Reference ID/Investigator# 8093, Paducah, Kentucky
  - Site Reference ID/Investigator# 38405, Baton Rouge, Louisiana
  - Site Reference ID/Investigator# 8903, Shreveport, Louisiana
  - Site Reference ID/Investigator# 21805, Auburn, Maine
  - Site Reference ID/Investigator# 8092, Rockville, Maryland
  - Site Reference ID/Investigator# 8225, Fall River, Massachusetts
  - Site Reference ID/Investigator# 8407, Springfield, Massachusetts
  - Site Reference ID/Investigator# 8415, Royal Oak, Michigan
  - Site Reference ID/Investigator# 22222, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 8408, Olive Branch, Mississippi
  - Site Reference ID/Investigator# 22703, Berlin, New Jersey
  - Site Reference ID/Investigator# 22707, Elizabeth, New Jersey
  - Site Reference ID/Investigator# 22702, Hillsborough, New Jersey
  - Site Reference ID/Investigator# 8387, Flushing, New York
  - Site Reference ID/Investigator# 8177, Great Neck, New York
  - Site Reference ID/Investigator# 8146, Lake Success, New York
  - Site Reference ID/Investigator# 22427, Williamsville, New York
  - Site Reference ID/Investigator# 22481, Charlotte, North Carolina
  - Site Reference ID/Investigator# 22708, Charlotte, North Carolina
  - Site Reference ID/Investigator# 8434, Morehead City, North Carolina
  - Site Reference ID/Investigator# 8417, Cincinnati, Ohio
  - Site Reference ID/Investigator# 8147, Columbus, Ohio
  - Site Reference ID/Investigator# 22488, Mason, Ohio
  - Site Reference ID/Investigator# 22479, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 23225, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 22482, Tulsa, Oklahoma
  - Site Reference ID/Investigator# 8345, Bend, Oregon
  - Site Reference ID/Investigator# 22704, Medford, Oregon
  - Site Reference ID/Investigator# 8400, Portland, Oregon
  - Site Reference ID/Investigator# 8411, Bethlehem, Pennsylvania
  - Site Reference ID/Investigator# 8405, Carlisle, Pennsylvania
  - Site Reference ID/Investigator# 22387, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 22815, Jersey Shore, Pennsylvania
  - Site Reference ID/Investigator# 12881, Johnstown, Pennsylvania
  - Site Reference ID/Investigator# 22706, Perkasie, Pennsylvania
  - Site Reference ID/Investigator# 8095, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 22705, Tipton, Pennsylvania
  - Site Reference ID/Investigator# 22817, Warminster, Pennsylvania
  - Site Reference ID/Investigator# 8098, Providence, Rhode Island
  - Site Reference ID/Investigator# 22823, Charleston, South Carolina
  - Site Reference ID/Investigator# 8364, Columbia, South Carolina
  - Site Reference ID/Investigator# 22429, Greenville, South Carolina
  - Site Reference ID/Investigator# 22428, Mt. Pleasant, South Carolina
  - Site Reference ID/Investigator# 25302, Summerville, South Carolina
  - Site Reference ID/Investigator# 22812, Dallas, Texas
  - Site Reference ID/Investigator# 8536, Edinburg, Texas
  - Site Reference ID/Investigator# 22810, Fort Worth, Texas
  - Site Reference ID/Investigator# 24742, Houston, Texas
  - Site Reference ID/Investigator# 26722, Houston, Texas
  - Site Reference ID/Investigator# 8406, Houston, Texas
  - Site Reference ID/Investigator# 8232, Lubbock, Texas
  - Site Reference ID/Investigator# 22480, San Antonio, Texas
  - Site Reference ID/Investigator# 8397, San Antonio, Texas
  - Site Reference ID/Investigator# 21804, Ogden, Utah
  - Site Reference ID/Investigator# 22423, Salt Lake City, Utah
  - Site Reference ID/Investigator# 8413, Gig Harbor, Washington
- Puerto Rico (12):
  - Site Reference ID/Investigator# 24402, Carolina
  - Site Reference ID/Investigator# 22545, Humacao
  - Site Reference ID/Investigator# 8301, Manatí
  - Site Reference ID/Investigator# 8299, Ponce
  - Site Reference ID/Investigator# 8418, Ponce
  - Site Reference ID/Investigator# 8419, Ponce
  - Site Reference ID/Investigator# 8421, San Juan
  - Site Reference ID/Investigator# 8300, San Juan
  - Site Reference ID/Investigator# 8422, San Juan
  - Site Reference ID/Investigator# 8423, San Juan
  - Site Reference ID/Investigator# 8420, Toa Baja
  - Site Reference ID/Investigator# 8298, Yabucoa

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Weinstein DL, Williams LA, Carlson DM, Kelly MT, Burns KM, Setze CM, Lele A, Stolzenbach JC. A randomized, double-blind study of fenofibric acid plus rosuvastatin compared with rosuvastatin alone in stage 3 chronic kidney disease. Clin Ther. 2013 Aug;35(8):1186-98. doi: 10.1016/j.clinthera.2013.06.013. Epub 2013 Jul 26. PMID 23891363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 280 participants were randomized and treated at 84 sites in the United States and Puerto Rico between 23 July 2008 and 02 March 2011.
Period: Overall Study
Arm/Group | ABT-335 Plus Rosuvastatin | Rosuvastatin
Started | 140 | 140
Completed | 123 | 128
Not Completed | 17 | 12
Not completed — Adverse Event | 13 | 7
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 Plus Rosuvastatin | Rosuvastatin | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 48 | 115
  >=65 years | 73 | 92 | 165
Age Continuous [Mean (Standard Deviation); unit: years] | 65.1 (10.35) | 67.4 (11.15) | 66.2 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 71 | 149
  Male | 62 | 69 | 131
Region of Enrollment [Number; unit: participants]
  United States | 129 | 132 | 261
  Puerto Rico | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change in Triglycerides From Baseline to Week 8.
Description: Triglycerides were measured in milligrams/deciliter.
Time Frame: Baseline to 8 weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 postbaseline value for triglycerides. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | ABT-335 Plus Rosuvastatin | Rosuvastatin
Number analyzed (Participants) | 137 | 138
percent change | -38.0 [-53.1 to -23.8] | -22.4 [-38.2 to -4.5]
Statistical Analysis 1: Comparison: ABT-335 Plus Rosuvastatin vs Rosuvastatin; The null hypothesis was that percent change in triglycerides (TG) from baseline to Week 8 in the ABT-335 45 mg plus rosuvastatin 5 mg treatment group is equal to percent change in TG from baseline to Week 8 in the rosuvastatin 5 mg plus placebo treatment group. A sample size of 140 participants per treatment group was used to provide 98% power to detect a difference between the combination therapy arm and the rosuvastatin monotherapy arm in the percent change from Baseline to Week 8 in TG; Test type: Superiority or Other; p < 0.001, Wilcoxon rank-sum test — P values were based on 2 sided tests. Tests resulting in P values less than or equal to 0.050 (when rounded) were reported as "statistically significant". No adjustments made for multiple comparisons since only 1 primary efficacy endpoint comparison

2. Secondary Outcome: Mean Percent Change in High-Density Lipoprotein Cholesterol From Baseline to Week 8.
Description: High-density lipoprotein cholesterol (HDL-C) was measured in milligrams/deciliter (mg/dL).
Time Frame: Baseline to 8 weeks
Population: Full Analysis Set was used and was defined as all randomized participants who had both a baseline value and at least 1 postbaseline value for HDL-C. Last observation carried forward (LOCF) was used to impute values for participants missing a post-baseline visit value. Only post-baseline values were carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | ABT-335 Plus Rosuvastatin | Rosuvastatin
Number analyzed (Participants) | 137 | 138
percent change | 16.9 (1.44) | 7.8 (1.43)
Statistical Analysis 1: Comparison: ABT-335 Plus Rosuvastatin vs Rosuvastatin; The null hypothesis was that percent change in HDL-C from baseline to Week 8 in the ABT-335 45 mg plus rosuvastatin 5 mg treatment group is equal to percent change in HDL-C from baseline to Week 8 in the rosuvastatin 5 mg plus placebo treatment group. A sample size of 140 participants per treatment group was used to provide 82% power to detect a difference between the combination therapy arm and the rosuvastatin monotherapy arm in the percent change from Baseline to Week 8 in HDL-C; Test type: Superiority or Other; p < 0.001, ANCOVA — P values were based on 2 sided tests. Tests resulting in P values less than or equal to 0.050 (when rounded) were reported as "statistically significant". No adjustments made for multiple comparisons since only 1 secondary endpoint comparison; P-value obtained from an ANCOVA with corresponding baseline value as the covariate and an effect for treatment group

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Treatment-emergent adverse events were defined as those occurring after study drug initiation and within 30 days after the last dose of study drug. Treatment-emergent serious adverse events were collected from the time the participant signed the informed consent until 30 calendar days following discontinuation of study drug.
Arm/Group | ABT-335 Plus Rosuvastatin | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 9/140 | 11/140
Other Adverse Events (participants affected / at risk) | 54/140 | 60/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 Plus Rosuvastatin (N=140) | Rosuvastatin (N=140)
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 3
Myocardial Infarction (Cardiac disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 Plus Rosuvastatin (N=140) | Rosuvastatin (N=140)
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 11
Vomiting (Gastrointestinal disorders) | 1 | 7
Fatigue (General disorders) | 0 | 10
Oedema Peripheral (General disorders) | 7 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 7
Blood Creatinine Increased (Investigations) | 8 | 2
Glomerular Filtration Rate Decreased (Investigations) | 12 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Headache (Nervous system disorders) | 5 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Hypertension (Vascular disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.